CLINICAL TRIAL: NCT00091884
Title: Efficacy of Elevated CD4 Cell Counts on CMV Retinitis
Brief Title: Efficacy of Elevated CD4 Counts on CMV Retinitis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040223; 04-EI-0223
Record Dates: First submitted 2004-09-17; First posted 2004-09-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis
Keywords: HIV; Immune Recovery; Reactivation; Anti-Viral Medication; HAART; CMV Retinitis; Retinal Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis; Retinal Diseases

SUMMARY:
Some patients with HIV/AIDS suffer from a dangerous viral infection of the retina (and other organs) called cytomegalovirus infection (CMV). The medications currently used to treat CMV all have serious side effects. AIDS patients are prone to this infection because their immune system produces a lower number of CD4+T lymphocytes, the type of blood cells that fight viral infections.

Some new HIV medications strengthen the immune system. This study will investigate the possibility that CMV patients on these HIV medications can develop immune systems strong enough to fight CMV without CMV medication. The study will enroll a maximum of 15 adult HIV/AIDS patients who have a CD4+T cell count over 150 cells/microliter and who have inactive CMV retinitis that is not immediately sight threatening. It is expected to last approximately 2 years.

Each prospective participant will have a physical examination and complete eye examination, including retina photographs, with the eye examination and retina photographs repeated 2 weeks later. If there is no evidence of active CMV retinitis, the participant will be enrolled in the study, and CMV medication will be stopped. The participant will have physical and eye examinations every 2 weeks for the first 3 months of the study, and every 3 weeks for the next 3 months. After 6 months, the frequency of the examinations will be 2-8 weeks, depending on the participant's CD4 count. After one year, a participant with a CD4 count remaining over 150 cells/microliter may return to the care of a local ophthalmologist with HIV/CMV experience, revisiting the clinical center every 6 months. The participant's CMV medication will be restarted when CMV retinitis becomes active, which will terminate participation in the study.

DETAILED DESCRIPTION:
This is a clinical trial to determine whether elevated CD4 counts resulting from medications against human immunodeficiency virus (HIV) are effective in controlling cytomegalovirus (CMV) retinitis. Patients with non-progressive retinal disease consistent with inactive CMV retinitis in a location that is not immediately sight threatening, who are currently receiving systemic maintenance therapy with ganciclovir, foscarnet, or cidofovir, and who have a total CD4 cell count greater than 150 cells per microliter will have their anti-CMV therapy discontinued. Patients will then be closely followed for progression of their CMV retinitis. The primary endpoint of the study will be progression of CMV retinitis. Secondary endpoints will include the occurrence of extraocular CMV disease, morbidity, mortality, virologic data, and HIV burden.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of AIDS as defined by the Centers for Disease Control.

Inactive, non-sight-threatening CMV retinitis. Non sight-threatening CMV retinitis is defined as CMV retinitis not within 1000 microns from the optic disc or 1000 microns from the fovea. Exception: patients with CMV retinitis within 1000 microns of the fovea or disc in only one eye, if visual acuity in that eye is worse than 20/400 without the use of eccentric fixation, and visual acuity in the other eye is 20/400 or better.

CD4 T cell count greater than 150 cells per microliter.

Patients must be able understand the nature of the study, agree to the provision, and understand and sign the informed consent form.

Women and men age 18 or older are eligible for enrollment.

Platelets greater than 25,000/microliter.

Hemoglobin greater than 8.5 gms.

Total neutrophil count greater than 750/mm(3).

Karnofsky performance score greater than or equal to 60.

Receiving systemic anti-CMV therapy.

Receiving anti-HIV therapy. If the patient is receiving IL-2, at least one month from last infusion must elapse prior to assessment for eligibility.

EXCLUSION CRITERIA:

Intraocular sustained release ganciclovir implant in the eye for less than 9 months, or other organ involvement from CMV infection requiring use of systemic ganciclovir or foscarnet.

CMV retinitis should not involve the retina solely anterior to the equator, or within 1000 microns from the optic disc, or within 1000 microns from the fovea. Exception: patients with lesions that have involved the fovea or disc and caused visual acuity worse than 20/400 without the use of eccentric fixation, may be included.

Opacification of the cornea, lens, or vitreous in either eye that precludes examination of the fundus.

Other retinal disease that could obscure the diagnosis of CMV retinitis, such as ocular toxoplasmosis.

Significant psychiatric or emotional disorders that would impair patient understanding or participation in the trial.

Life expectancy less than three months.

Active CMV disease requiring systemic anti-CMV therapy.

CMV retinitis first diagnosised with CD4 T-cell count greater than 150 cells per microliter.

Need for medications with anti-CMV effect.

Participation in conflicting clinical trial.

Progression of CMV retinitis between screening and baseline examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2004-07; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Guarda LA, Luna MA, Smith JL Jr, Mansell PW, Gyorkey F, Roca AN. Acquired immune deficiency syndrome: postmortem findings. Am J Clin Pathol. 1984 May;81(5):549-57. doi: 10.1093/ajcp/81.5.549. PMID 6326563
- [Background] Moskowitz L, Hensley GT, Chan JC, Adams K. Immediate causes of death in acquired immunodeficiency syndrome. Arch Pathol Lab Med. 1985 Aug;109(8):735-8. PMID 2990379
- [Background] Palestine AG, Rodrigues MM, Macher AM, Chan CC, Lane HC, Fauci AS, Masur H, Longo D, Reichert CM, Steis R, et al. Ophthalmic involvement in acquired immunodeficiency syndrome. Ophthalmology. 1984 Sep;91(9):1092-9. doi: 10.1016/s0161-6420(84)34201-4. PMID 6093020